CLINICAL TRIAL: NCT02815163
Title: The Effects of Using the Empowerment Model Intervention in Primary Total Hip
Brief Title: The Effects of Using the Empowerment Model Intervention in Primary Total Hip Replacement Surgery Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tzu-Ting Huang (Other)
Responsible Party: Sponsor-Investigator, Tzu-Ting Huang, Professor, School of Nursing, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 97-2081B
Record Dates: First submitted 2016-06-21; First posted 2016-06-28 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Empowerment
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- comparison group (No Intervention): The CG received no extra care; they could receive the usual routine care for THR in the unit as they had before participation in the study. The routine care included oral instruction by nurses follow by the handout. Also, a brochure was provided of the structure of hip, the risk factors of THR, care before and after THR, complications, care of discharge, and demonstration of rehabilitation with pictures) of THR designed by researchers in this study. Five orthopedics health care experts independently reviewed and rated each item in the brochure on a five-point Likert-type scale in terms of relevance, representativeness, specificity, and clarity.
- Empowerment education group (Experimental): The 5 times total, 12-week EE intervention was aimed to empower older patients with THR to develop their own self-management program to meet their needs. This empowerment education intervention based on 6 empowerment components: "Partnership, listening, dialogue, reflection, action, feedback" and 5-step empowerment strategies: motivating patients self-awareness, assessing the causes of the problem, goal setting, individual self-care plan development, and checking whether goals or plans have been achieved who modified from Freire's 3-stage methodology. The difference between this program and the other health educations for patients with THR are that this program encourages them to explore their needs and worries, their own ability and power to meet their needs, and their capacity to seek and use their social support and resources etc.
  Interventions: Other: Empowerment education

INTERVENTIONS:
Other: Empowerment education — 1. admission (1 hour)
     ▪partnership
  2. 2 ds after THR (30-45min)
     * listening
     * dialogue
     * reflection
     * action
     * feedback
  3. 2 WKs after THR (30 min)
     * listening
     * dialogue
     * reflection
     * action
     * feedback
  4. 6 WKs after THR (30 min)
     * listening
     * dialogue
     * reflection
     * action
     * feedback
  5. 10 WKs after THR (30 min)
     * listening
     * dialogue
     * reflection
     * action
     * feedback
  Arms: Empowerment education group

SUMMARY:
Degenerative arthritis is a common and serious chronic illness that impacts the quality of life of older adults. Knowledge about the effects of empowerment education program in older adults with total hip replacement surgery are limited. As far as the investigators know, this is the first study done using empowerment education intervention to promote total hip replacement patients' self-care. This partnership is achieved through active participation to learn as well as sharing their knowledge and experiences with clinicians and patients. Furthermore, patients had developed some degree of self-efficacy and improve their depressive mood from the disease related knowledge acquired.

DETAILED DESCRIPTION:
Aims. To exam the effectiveness of the empowerment education program on primary (self-care self-efficacy and competence) and secondary outcomes (Activities of Daily Life, mobility, depressive mood, and quality of life) for older adults with total hip replacement surgery.

Background. Degenerative arthritis is a common and serious chronic illness that impacts the quality of life of older adults. As joints degenerate continuously and the hip has been damaged by arthritis, Activities of Daily Life will be difficult to perform due to severe hip pain and joint stiffness. Therefore, hip replacement surgery should be considered, and effective nursing care should be provided to improve the recovery of older adults.

Design. A prospective randomized control trial. Methods. A trial was conducted from September of 2013 to May of 2014 in two hospitals in northern Taiwan. 108 participants were randomly assigned to either the empowerment education group or the comparison group. The outcomes were collected at the day of discharge (T2), one month after (T3), and 3 months (T4) after the discharge.

ELIGIBILITY:
Inclusion Criteria:

* had 1st THRS
* ability to speak and read Chinese
* willingness to participate in this study

Exclusion Criteria:

* cognitive impairment or been diagnosed with a psychiatric illness
* participation in another study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Total Hip Replacement Self-efficacy Scale | 5min
  A five-item evaluation list measured self-efficacy (environment, self-monitoring, regular check-up, medicine, exercise), all components were rated on a 5-point Likert-type scale (4= fully confident to 0= no confidence at all) with higher scores signifying greater self-efficacy.
Self-care competence Scale | 5min
  The knowledge and behaviors subscales measured this variable, which includes knowledge and behavior related to THR self-care. The knowledge subscale contains 15 yes/no questions (6 for posture/ environment, 6 for wound/pain, and 3 for exercise), each with only one correct response. In order to prevent participants that guessed answers from confounding the data, the choice 'I do not know' was also provided. The scores range from 0 to 15, with higher scores indicating greater knowledge.

SECONDARY OUTCOMES:
ADL | 3min
  ADL was assessed using the Barthel scale, which was introduced in 1965 and yielded a score of 0-100, the measure 10 variables. These variables included fecal incontinence, urinary incontinence, and assistance with grooming, feeding, transfers, walking, dressing, climbing stairs, and bathing.
Tinetti mobility | 3min
  The Tinetti Mobility Scale (Tinetti et al. 1986) assessed mobility (gait and balance). This scale is simple: no required equipment attached and is quick and convenient to use. Each participant took around 5 minutes to perform the series of activities to assess mobility. The better a participant's performance, the higher the score.
GDS-15 | 3min
  consisting of 15 questions, was the primary outcome evaluator (Sheikh and Yesavage, 1986). Scores of 0-4 are considered to be normal; 5-8 indicates mild depression; 9-11 indicates moderate depression; and 12-15 indicates severe depression.
SF-36 | 3min
  The SF-36 questionnaire assesses health-related functions for eight distinct domains, which can be divided into physical component and mental component scales. This 36-item questionnaire was used to measure quality of life.

IPD SHARING:
Plan to Share IPD: No